CLINICAL TRIAL: NCT03139396
Title: Clinical Assessment Of Inlay Retained Bridge Designs (Tub Shaped And Inlay Shaped) In Missing Posterior Teeth Cases. (Randomized Clinical Trial)
Brief Title: Assessment Of Inlay Retained Bridge Designs In Missing Posterior Teeth Cases. (Randomized Clinical Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Abdelgawad, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-04-16
Record Dates: First submitted 2017-04-30; First posted 2017-05-04 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Tooth Loss
Keywords: inlay bridge, tub shaped design
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inlay shaped inlay bridge design (Active Comparator): The inlay shaped inlay bridge design preparation show three types of preparation, the inlay shaped, the tub shaped inlay bridge design and the proximal box shaped designs. Intracoronal preparation of the inlay retained prosthesis for the abutments (inlay shaped and tub shaped) should show the following criteria: The inlay shaped preparation should show an occlusal-proximal box preparation and to be designed with the line angles should be rounded, smooth and rounded corners, and rectangular flat floor with no beveling for the occlusal and gingival margins. The occlusal inlay preparation should have preparation depth allowed for a thickness of 2.0 mm for the material of the bridge. The occlusal reduction show 4 mm width with extension of 4 or 6 mm mesio distally for the posterior teeth.
  Interventions: Procedure: tub shaped inlay bridge design
- tub shaped inlay bridge design (Experimental): The tub-shaped reduction consist of an occlusal proximal inlay and prepared as the same geometry as the inlay shaped preparation, except that for the proximal box preparation which is not present in this preparation design.
  Interventions: Procedure: tub shaped inlay bridge design

INTERVENTIONS:
Procedure: tub shaped inlay bridge design — inlay retained bridge with tub shaped retainer on both abutments
  Other Names: tub shaped

SUMMARY:
Patients with missing back teeth can be restored with an inlay retained bridge.The inlay retained bridge designs include inlay shaped, tub shaped or proximal box shaped.In this study a clinical evaluation will be commenced to evaluate two designs the inlay shaped and the tub shaped.The hypothesis of our trial is that the new design may show longer survival rate due to less stress applied on the restoration which allow the restoration to function for longer period as the inlay shaped bridge showed clinical problems during survice.

DETAILED DESCRIPTION:
: This trial will be conducted on patients from the Outpatient clinic in the Fixed Prosthodontics Clinic, Faculty of Oral and Dental Medicine, Cairo University.

- Adherence session will take place in the presence of the patients in the initial visit. This include that the patient will be informed by Abdelfattah M about the study steps and maintenance of oral hygiene instructions. Participants will be asked by Abdelfattah M about if they have any problems like pain.

Motivation and enforcing the maintenance of oral hygiene measures by Abdelfattah M.

The visits will be designated as follows:

Visit 1: Preoperative records, face-to-face adherence reminder session, clinical examination, radiographic examination, intraoral photography and primary impressions (Zhermack ) for diagnostic cast construction ( Zhermack ) . Visit 2: teeth preparations, secondary impression ( Zhermack ) and temporization (Tempofit) .

Visit 3: try in for the restoration. Visit 4: final cementation of the restoration.(GC resin cement) Visit 5: follow up

Sample size:

As there is no previously published effect size data regarding the effectiveness of the intervention or the control, an estimated sample size of 10 bridges would be used with allocation ratio of 1:1.

Recruitment:

The patients who show the inclusion criteria as mentioned will be selected by Abdelfattah M from the outpatient clinic of the fixed prosthodontics department - Cairo University. Screening will be carried out by Abdelfattah M for patients until the target population is reached.

Methods: Assignment of interventions:

Sequence generation The participant will be allocated in to two groups with 1:1 allocation ratio by using computer by Abdelfattah M.

Implementation:

Abdelfattah (the main researcher) will select the patients who show the listed inclusion criteria and divided them into two groups Blinding An independent examiner (not the main researches) will assess the all restorations (double blind study).

Plans to promote participant retention & complete follow-up:

Telephone numbers and addresses of the patients enrolled in the trial will be recorded by Abdelfattah M. All patients will be given a phone call before the next appointment for confirming to their coming. Efforts will be done to achieve proper participant retention like explaining the next procedure to the participant, elaborate to the participants the benefits gained from being enrolled in the study and use a schedule for the next visits.

Data management All data will be managed electronically. Patient files will be stored in numerical order in a secured place. This will be carried out by Abdelfattah M Data analysis All Data will be collected, revised, arranged in tables and entered into the system by Abdelfattah M. Quantitative variables from normal distribution will be expressed as mean and standard deviation (SD) values. To test the significant differences between two groups student t-test will be used. Significant level will be set at P ≤ 0.05. Statistical analysis will be done using Statistical Package for Social Sciences, Version 21.0 (SPSS, IBM, Chicago, III, USA) for Windows.

Data monitoring Data monitoring is the responsibility for the main supervisor (El Mahallawi O). Interim analysis will be done if harms occur.

Harms Any harm or adverse events like pain or failure if happened will be recorded, documented and dealed with as recommended by Abdelfattah M.

Consent Abdelfattah M will discuss all study aspects with all patients, so patients will be able to have an informed discussion with the researcher. Abdelfattah M will obtain written consent from the patients who willing to participate in the study. All consent forms will be in Arabic language Confidentiality All information related to the study will be stored in a secure place. All patients information will be stored in cabinets in areas with limited access. All data processing forms will be identified by a number to maintain participant confidentiality.

Access to data Access to the data is allowed to the investigator and supervisors. The participant study information will be confidential.

Ancillary care All patients will be followed up until the study period is completed. As any prosthetic treatment, post insertion adjustments will be done if necessary and the recall maintenance visits will be arranged.

Dissemination policy

* The results of the study will be published as partial fulfillments for the doctorate degree in fixed prosthodontics.
* Topics from the study suggested for presentation or publication will be circulated to the authors.

Data collection:

Primary outcome: the retention of the restoration for both groups will be assessed using MUSPHS criteria.

Secondary outcome: the marginal fit, caries, fracture and gingivitis for both groups will be assessed using the MUSPHS and gingival index.

ELIGIBILITY:
Inclusion Criteria:

1. From 18-55 years old, should be able to read and sign the consent document.
2. Ability to tolerate the restorative procedures (physical and psychological).
3. Patients with teeth problems indicated for inlay retained fixed partial denture:

   1. Good oral hygiene
   2. Low susceptibility to decay
   3. Have a minimum coronal tooth height of 5 mm,
   4. Parallel abutments
   5. Sufficient mesio distal edentulous gap dimensions.
4. With no active periodontal or pulpal problems, with sound teeth or teeth with shallow restorations
5. Willing to return for follow-up visits.

Exclusion Criteria:

1. Partially erupted teeth (young)
2. Bad oral hygiene and motivation
3. Root canal treated teeth
4. Psychiatric problems or unrealistic expectations
5. Severe parafunctional habits
6. The absence of enamel on the preparation margins
7. Extensive crown defects
8. Abutment mobility

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Retention | 1 year
  assess the loss of the restoration (debonding) the scale that will be used is the MUSPHS scale and the measuring unit is score (discrete)

SECONDARY OUTCOMES:
marginal adaptation | 1 year
  assess the fitting of the restoration on the underlying tooth the scale that will be used is the MUSPHS scale and the measuring unit is score (discrete)
Caries | 1 year
  assess if decay occurred on the abutment teeth the scale that will be used is the MUSPHS scale and the measuring unit is score (discrete)
gingivitis | 1 year
  assess if the gum aroung the teeth is inflamed the scale that will be used is the Gingival index scale and the measuring unit is score (discrete)
fracture | 1 year
  assess if cracks or fracture occurred to the restoration the scale that will be used is the MUSPHS scale and the measuring unit is score (discrete)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Izgi AD, Kale E, Eskimez S. A prospective cohort study on cast-metal slot-retained resin-bonded fixed dental prostheses in single missing first molar cases: results after up to 7.5 years. J Adhes Dent. 2013 Feb;15(1):73-84. doi: 10.3290/j.jad.a29010. PMID 23534027
- [Background] Ohlmann B, Rammelsberg P, Schmitter M, Schwarz S, Gabbert O. All-ceramic inlay-retained fixed partial dentures: preliminary results from a clinical study. J Dent. 2008 Sep;36(9):692-6. doi: 10.1016/j.jdent.2008.04.017. Epub 2008 Jun 11. PMID 18550253